CLINICAL TRIAL: NCT00022555
Title: A Phase I Trial of Combination Bryostatin-1 and Vincristine in HIV-Related B-cell Neoplasms
Brief Title: Bryostatin 1 Plus Vincristine in Treating Patients With Recurrent or Refractory HIV-Related Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02398; AMC-029; U01CA070019 (NIH); CDR0000068830 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Diffuse Mixed Cell Lymphoma; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Small Noncleaved Cell Lymphoma
MeSH Terms: interventions — bryostatin 1; Bryostatins; Vincristine

ARMS (1):
- Treatment (bryostatin 1, vincristine sulfate) (Experimental): Patients receive bryostatin 1 IV continuously on days 1 and 15 and vincristine IV over 5 minutes on days 2 and 16. Treatment continues every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bryostatin 1; Drug: vincristine sulfate

INTERVENTIONS:
Drug: bryostatin 1 — Given IV
  Other Names: B705008K112; BRYO; Bryostatin
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS

SUMMARY:
Phase I trial to study the effectiveness of bryostatin 1 plus vincristine in treating patients who have recurrent or refractory lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Bryostatin 1 may help vincristine kill more cancer cells by making them more sensitive to the drug

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of bryostatin 1 when administered with vincristine in patients with recurrent or refractory HIV-related B-cell lymphoma.

II. Determine the toxicity profile of this regimen in these patients. III. Determine the objective response and survival of these patients treated with this regimen.

IV. Determine the immunomodulatory effects of this regimen on interleukin-2 (IL-2), IL-2 receptor, and IL-6 cytokine levels in these patients.

V. Determine the effect of this regimen on CD4+ lymphocyte count and HIV load in these patients.

VI. Determine the effect of this regimen on the human herpes virus-8 load in these patients with body cavity-based lymphoma.

OUTLINE: This is a multicenter, dose-escalation study of bryostatin 1.

Patients receive bryostatin 1 IV continuously on days 1 and 15 and vincristine IV over 5 minutes on days 2 and 16. Treatment continues every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bryostatin 1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell lymphoma

  * Eligible subtypes:

    * Intermediate or high-grade non-Hodgkin's lymphoma (NHL), defined as follicular large cell, mantle cell, diffuse mixed cell, diffuse large cell and variants, Burkitt or Burkitt-like, or unclassifiable aggressive histologies
    * Body cavity-based lymphoma or primary effusion lymphoma
* Evidence of HIV infection
* Received at least 1 prior systemic chemotherapy regimen with failure to respond or relapse after completion of first-line therapy, including one of the following doxorubicin-based combinations:

  * Cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP)
  * Infusional cyclophosphamide, doxorubicin, and etoposide (CDE)
  * Etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (EPOCH)
* Evaluable disease outside of prior radiation port
* No CNS parenchymal or leptomeningeal involvement
* No primary CNS NHL
* No HTLV-1-associated leukemia or lymphoma
* Performance status - Karnofsky 70-100%
* At least 12 weeks
* Absolute granulocyte count at least 1,000/mm3
* Platelet count at least 75,000/mm3
* Hemoglobin at least 8.0 g/dL
* Bilirubin no greater than 1.5 mg/dL (unless concurrently on indinavir)
* SGOT and SGPT less than 3 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 50 mL/min
* No history of cardiac disease
* LVEF at least 45% by radionuclide ventriculography
* No symptomatic congestive heart failure
* No active angina pectoris
* No uncontrolled hypertension
* No history of symptomatic pulmonary disease
* Corrected DLCO more than 50% predicted
* No severe chronic obstructive lung disease
* No symptomatic restrictive lung disease
* Recurrent controllable infection (e.g., thrush) on chronic suppressive therapy allowed
* No active uncontrolled infection
* No active significant opportunistic infection (e.g., acute Pneumocystis pneumonia, cytomegalovirus retinitis on induction or maintenance therapy, acute toxoplasmosis)
* No grade 2 or greater peripheral neuropathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* At least 24 hours since prior transfusion
* At least 24 hours since prior colony-stimulating factor therapy
* No concurrent prophylactic filgrastim (G-CSF)
* See Disease Characteristics
* No concurrent hydroxyurea
* See Disease Characteristics
* At least 4 weeks since prior large-field radiotherapy
* At least 3 weeks since prior anticancer therapy and recovered
* Must be receiving stable antiretroviral regimen of at least 4 weeks duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-11; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
MTD of bryostatin-1 defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity | 4 weeks

SECONDARY OUTCOMES:
Dose-limiting toxicities | 4 weeks
  Defined as any >= grade 2 neuropathy, other grade 3 non-hematologic toxicity (excluding alopecia and grade 3 nausea and vomiting that is responsive to standard pharmacologic intervention) or grade 4 hematologic toxicity in 2 or more patients. The incidence of toxicity related dose reduction and treatment discontinuation will be summarized for each dose group.
Immunomodulatory effects of this combination | Up to 2 years
  Measured by a solid phase Enzyme Amplified Sensitivity Immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Scot Remick, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (1):
- AIDS - Associated Malignancies Clinical Trials Consortium, Rockville, Maryland, United States